CLINICAL TRIAL: NCT04194424
Title: A Multidisciplinary Weight Loss Program at AUB-MC: An Open Label Pilot Randomized Controlled Trial
Brief Title: A Multidisciplinary Weight Loss Program at AUB-MC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Marlene Chakhtoura, Assistant Professor of Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2018-0400
Record Dates: First submitted 2019-07-18; First posted 2019-12-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Standard of Care; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidisciplinary program (Experimental): Multidisciplinary weight loss program
  Interventions: Other: Multidisciplinary weight loss program; Drug: Metformin Hcl 850Mg Tab
- Control (Other): Standard care
  Interventions: Other: Standard Care; Drug: Metformin Hcl 850Mg Tab

INTERVENTIONS:
Other: Multidisciplinary weight loss program — Diet and behavioral therapy,and supervised exercise sessions
  Arms: Multidisciplinary program
Other: Standard Care — General lifestyle tips
  Arms: Control
Drug: Metformin Hcl 850Mg Tab — 1 tablet, twice daily

SUMMARY:
The current project aims at evaluating the feasibility and efficacy of a multi-disciplinary weight loss program, using an innovative and simple dietary intervention at the American University of Beirut Medical Center (AUB-MC). Such intervention is expected to enhance patients' compliance and adherence to lifestyle changes. In addition, the program includes supervised exercise sessions and behavioral therapy. Therefore, our project proposes an evidence based approach to close the obesity treatment gaps.

ELIGIBILITY:
Inclusion Criteria:

* Lebanese adult with obesity (≥18 years), obesity being defined as BMI ≥ 30 kg/m2
* Patients who can commit to frequent visit trials as per study protocol
* Patients not traveling outside Lebanon for at least the 6-month period of the trial
* Patients tolerating Metformin after a run-in period of 2 weeks

Exclusion Criteria:

* Patients who have taken other weight reducing drug therapy in the previous 6 months
* Patients who have undergone bariatric therapy or endoscopic procedure, or planning to do so in the near future (at < 6 months)
* Patients with diabetes
* Patients working at AUB-MC, as we will not be able to assess the adherence to study visits nor the feasibility of such a program in the general population, presenting to AUB-MC only for clinical care
* A family member of a patient already enrolled in the study, as the participants will not be independent
* Pregnant obese patients
* Patients with pacemakers
* Patients known to have hypertension, cardiac, pulmonary, renal or liver disease, active cancer or psychiatric illnesses
* History of any surgery of less than 6 weeks duration
* Patients known to have disabling osteoarthritic or orthopedic problems
* Patients secondary uncontrolled endocrine disorders (thyroid disorders, polycystic ovary, Cushing disease), or drug induced obesity (such as anti-psychotic, steroids, hormonal therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Mean percent weight loss per treatment arm | 6 months after enrollment
  [(baseline weight-follow up weight at 6 months)/ baseline weight] X 100

OTHER OUTCOMES:
Change in weight | 6 months after enrollment
  TANITA Body Composition (BC) 418 MA Segmental Body Composition Analyzer will measure Weight in kg
Change in BMI | 6 months after enrollment
  TANITA BC 418 MA Segmental Body Composition Analyzer will measure BMI (kg/m^2) by combining the height and weight.
Change in body composition | 6 months after enrollment
  TANITA BC 418 MA Segmental Body Composition Analyzer will measure total body measurements for: Fat Mass, Fat Free Mass, Total Body Water (in kg)
basal metabolic rate (BMR) | 6 months after enrollment
  TANITA BC 418 MA Segmental Body Composition Analyzer will measure BMR
Change in physical fitness (distance) | 6 months after enrollment
  Physical fitness will be assessed using the 6 minute walk test. Measure to be collected at beginning and end of test is: distance covered in meters
Change in resting blood pressure before and after physical exercise | 6 months after enrollment
  Physical fitness will be assessed using the 6 minute walk test. Measure to be collected at beginning and end of test is: resting blood pressure
Change in oxygen saturation before and after physical exercise | 6 months after enrollment
  Physical fitness will be assessed using the 6 minute walk test. Measure to be collected at beginning and end of test is: oxygen saturation
Change in heart rate before and after physical exercise | 6 months after enrollment
  Physical fitness will be assessed using the 6 minute walk test. Measure to be collected at beginning and end of test is: heart rate.
Change in physical fitness (Perceived Exertion) | 6 months after enrollment
  Physical fitness will be assessed using the 6 minute walk test. Rated Perceived Exertion (RPE) scale score will be administered.
Change in levels of appetite hormones and metabolic markers | 6 months after enrollment
  At visit 3 and completion visit (visit 5), blood samples will be withdrawn for various hormones and proteins related to appetite and satiety including Gastric inhibitory polypeptide (GIP), Leptin, Glucagon like peptide 1 (GLP1), Irisin, Insulin, Ghrelin, Orexin, IL6
  These samples will be processed and preserved in the Calcium Metabolism and Osteoporosis Program lab in our institution, and the tests will be run later on, when additional funds are available.
Change in levels of Mineral markers and hormones (cross laps) | 6 months after enrollment
  At visit 3 and completion visit (visit 5), blood samples will be withdrawn for various mineral markers and hormones including Crosslaps (pg/mL).
  These samples will be processed and preserved in the Calcium Metabolism and Osteoporosis Program lab in our institution, and the tests will be run later on, when additional funds are available.
Change in levels of Mineral markers and hormones (Osteocalcin) | 6 months after enrollment
  At visit 3 and completion visit (visit 5), blood samples will be withdrawn for various mineral markers and hormones including Osteocalcin (ng/mL).
  These samples will be processed and preserved in the Calcium Metabolism and Osteoporosis Program lab in our institution, and the tests will be run later on, when additional funds are available.
Participants' compliance | 6 months after enrollment
  Adherence to the dietary intervention: [Number of days the dieticians are contacted/ Total number of days] X 100 Adherence to program visits: [Number of visits attended/ Total number of visits] X 100

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut - Medical Center, Beirut, Riad El Solh, Lebanon

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT04194424/Prot_SAP_000.pdf